CLINICAL TRIAL: NCT06390579
Title: Building Research With Artificial Intelligence in Neuro-Ophthalmology
Acronym: BRAIN
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20230926_8_DMA_BRAIN
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Optic Neuropathy; Optic Neuropathy, Ischemic; Optic Neuritis; Optic Nerve Diseases; Papilledema; Optic Atrophy; Brain Tumors; Retinal Photograph; Artificial Intelligence (AI); Machine Learning; Deep Learning
Keywords: fundus imaging; automated diagnosis; multi-class classification; clinical decision support
MeSH Terms: conditions — Optic Nerve Diseases; Optic Neuropathy, Ischemic; Optic Neuritis; Papilledema; Optic Atrophy; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Deep learning algorithm applied on retrospectively collected color fundus photographs — Deep learning algorithm applied on retrospectively collected color fundus photographs

SUMMARY:
The research team, recognized as a world leader in Artificial Intelligence for neuro-ophthalmology, has shown that it is possible to diagnose certain neuro-ophthalmologic or neurologic disorders from a single retinal fundus image (Milea et al, New England Journal of Medicine, 2020). However, clinical practice requires identifying a broader spectrum of diseases (inflammatory, ischemic, hereditary, neurodegenerative) within the same analysis.

The main objective is to develop, through a new algorithm capable of classifying multiple disorders from a smaller set of conventional retinal images.

This project meets a significant public health need: the global shortage of neuro-ophthalmologists. It aims to provide healthcare professionals with a rapid triage tool to detect serious and treatable conditions, enabling timely intervention.

The study will include patients with clearly defined neuro-ophthalmologic or neurologic conditions, confirmed diagnoses, and retinal imaging. Clinical, paraclinical, and imaging data collected during standard care will be used, with strict anonymization according to legal and institutional requirements.

Specific Objectives :

1. Evaluate the performance of a diagnostic classification algorithm trained on retinal images.
2. Assess the ability to detect multiple pathologies from a single retinal image.
3. Support the development of advanced computer vision tools for medical diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-defined neuro-ophthalmologic or neurologic conditions, including different forms of optic neuropathies and various neurodegenerative diseases.
* Patients with a robust reference diagnosis confirmed by clinical experts.
* Patients with available retinal fundus images collected during routine care.

Exclusion Criteria:

* Patients without a confirmed diagnosis or unclear clinical classification.
* Patients without retinal fundus images or with images that are completely unreadable.
* Patients whose data cannot be anonymized according to legal and institutional protocols.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Color fundus photographs taken within 30 days from the date of onset
Sampling Method: Non-Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the Artificial Intelligence algorithm in detecting multiple neuro-ophthalmologic and neurologic conditions from retinal imaging. | baseline
  Evaluation of the algorithm's sensitivity, specificity, and area under the receiver operating caracteristics curve for classifying multiple neuro-ophthalmologic and neurologic pathologies using retinal fundus photography and Optical Coherence Tomography images, compared with expert-established reference diagnoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gungor A, Sarbout I, Gilbert AL, Hamann S, Lebranchu P, Hobeanu C, Gohier P, Vignal-Clermont C, Dumitrascu OM, Cohen SY, Lagreze WA, Feltgen N, van der Heide F, Lamirel C, Jonas JB, Obadia M, Racoceanu D, Milea D. Artificial Intelligence-Based Detection of Central Retinal Artery Occlusion Within 4.5 Hours on Standard Fundus Photographs. J Am Heart Assoc. 2025 Jul;14(13):e041441. doi: 10.1161/JAHA.124.041441. Epub 2025 Jun 27. PMID 40576025